CLINICAL TRIAL: NCT00667082
Title: NPI-0052 and Vorinostat in Patients With Non-small Cell Lung Cancer, Pancreatic Cancer, Melanoma or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NPI-0052-103
Record Dates: First submitted 2008-04-22; First posted 2008-04-25 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Non-Small Cell Lung Cancer; Pancreatic Cancer; Melanoma; Lymphoma; Multiple Myeloma
Keywords: Non small Cell Lung Cancer; Pancreatic Cancer; Melanoma; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Melanoma; Lymphoma; Multiple Myeloma | interventions — marizomib; Vorinostat; Proteasome Inhibitors; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPI-0052 + Vorinostat Dose-Escalation (Experimental): 4 dose-escalation cohorts
  Interventions: Drug: NPI-0052 (marizomib) + vorinostat

INTERVENTIONS:
Drug: NPI-0052 (marizomib) + vorinostat — NPI-0052 IV injection over 1 to 10 minutes at doses ranging from 0.15 to 0.7 mg/m2 on Days 1, 8, and 15 of each 28-day Cycle
  Oral vorinostat 300 mg was administered with food on Days 1 to 16 of each 28-day Cycle
  Other Names: marizomib; proteasome inhibitor; HDAC inhibitor; Zolinza

SUMMARY:
This is a clinical trial examining the safety, pharmacokinetics, pharmacodynamics and efficacy of IV NPI-0052 (a proteasome inhibitor) in combination with oral vorinostat (Zolinza; a HDAC inhibitor) in patients with non-small cell lung cancer, pancreatic cancer, melanoma or lymphoma. Proteasome inhibitors block the breakdown of proteins by cells and HDAC inhibitors block modification of proteins regulating gene expression in cells. Both of these actions preferentially affect cancer cells, and the combination of the two has been seen to have a greater effect in laboratory studies.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky Performance Status (KPS) at 70% or more.
2. Non-small cell lung cancer, pancreatic adenocarcinoma, melanoma or lymphoma for which a standard, approved therapy is not available. Patients must have lesions that are evaluable by RECIST criteria.
3. All Adverse Events of any prior chemotherapy, surgery, or radiotherapy, must have resolved to CTCAE (v. 3.0) Grade 1 or less(except for hemoglobin).
4. Adequate bone marrow, renal, liver function.
5. Signed informed consent.

Exclusion Criteria:

1. Recent administration of chemotherapy, biological, immunotherapy or investigational agent, major surgery, or radiotherapy.
2. Intrathecal therapy.
3. Known brain metastases.
4. Significant cardiac disease.
5. Prior treatment with vorinostat or NPI-0052, or other HDACi (including valproic acid) or proteasome inhibitors.
6. Known allergy to any component of vorinostat. Prior hypersensitivity reaction of CTCAE Grade > 3 to therapy containing propylene glycol or ethanol.
7. Pregnant or breast-feeding women.
8. Concurrent, active secondary malignancy for which the patient is receiving therapy.
9. Significant active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of the combination NPI-0052 and Vorinostat | continuously

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics and pharmacodynamics of NPI-0052 and vorinostat | continuous
To evaluate the safety and toxicity profile of the combination of NPI-0052 and vorinostat | continuous
To evaluate the anti-tumor activity of NPI-0052 and vorinostat | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Reich, MD, Study Director — Triphase Research and Development I Corp
Locations (3):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Sir Charles Gairdner Hospital and University of Western Australia, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided